CLINICAL TRIAL: NCT01863381
Title: Comparison of Continuous Non-Invasive and Invasive Intracranial Pressure Measurement: Continuous Intracranial Pressure Monitoring Subprotocol
Brief Title: Comparison of Continuous Non-Invasive and Invasive Intracranial Pressure Measurement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: LifeBridge Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMST02802
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Hydrocephalus; Idiopathic Intracranial Hypertension; Pseudotumor Cerebri
Keywords: Hydrocephalus; Idiopathic intracranial hypertension; Pseudotumor cerebri; ICP; Intracranial pressure; CSF pressure; VIIP
MeSH Terms: conditions — Hydrocephalus; Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocephalus/Pseudotumor (Experimental): Patients between the ages of 18-65 years with suspected hydrocephalus or idiopathic intracranial hypertension (IIH), also known as pseudotumor cerebri, who are recommended by their doctor based on standard clinical criteria to undergo intracranial pressure monitoring. The interventions include tympanic membrane displacement (TMD) and DPOAE.
  Interventions: Device: Tympanic membrane displacement (TMD); Device: DPOAE

INTERVENTIONS:
Device: Tympanic membrane displacement (TMD) — The CCFP Analyser has a passive mode and an active mode. When used in active mode, the device generates a tone burst that is transmitted to the ear to elicit contraction of the stapedius muscle. The passive mode requires no stimulus or sound burst.
  For the lying, sitting, standing, and 10-degree head-down tilt conditions, the active mode will be used. Each condition comprises 13 stimuli of 0.3s duration.
  Overnight recording of non-invasive ICP will be done using the passive mode of the CCFP device.
  Other Names: Cerebral and Cochlear Fluid Pressure Analyzer (CCFP); Marchbanks; CCFP
Device: DPOAE — DPOAE measurement uses a clinical acoustic probe to record the ear's response to two simultaneous tones. DPOAE measurements will be made for 13 tones. The total measurement time for each condition is 2-4 minutes.
  Other Names: Distortion Product Otoacoustic Emissions

SUMMARY:
This research is being done to determine the accuracy of two noninvasive methods of measuring the pressure of the cerebrospinal fluid (CSF), also known as intracranial pressure or ICP.

DETAILED DESCRIPTION:
Recently, astronauts in long-duration spaceflight have been found to have a syndrome consisting of swelling of the optic nerve, impaired vision, and elevated cerebrospinal fluid pressure (also known as intracranial pressure [ICP]) via lumbar puncture (LP), which is similar to the syndrome of idiopathic intracranial hypertension (IIH). In astronauts, this syndrome is called Visual Impairment/Intracranial Pressure (VIIP). It is not possible to perform an LP on astronauts in space. Noninvasive methods of estimating ICP exist but have not been tested against continuous ICP methods in a patient cohort that is physiologically similar to that of astronauts.

The primary objective of this study is to determine the validity, reliability, accuracy, and precision of two noninvasive methods of ICP measurement (tympanic membrane displacement (TMD, Marchbanks Measurements Systems, UK) and distortion product otoacoustic emissions (DPOAE) in comparison to a reference standard, invasive ICP measurement, in human subjects undergoing diagnostic ICP monitoring.

The two noninvasive methods are based on the responses of the inner ear and middle ear to changes in ICP. The first method is TMD, which measures tiny movements of the ear drum, and the second is DPOAE, which is routinely used for newborn hearing screening.

Adults with hydrocephalus or pseudotumor cerebri who have been recommended on the basis of standard clinical criteria to have ICP monitoring either by insertion of a temporary spinal catheter or by insertion of a needle into an existing shunt reservoir are eligible.

After insertion of the spinal catheter or the needle in the shunt, subjects will undergo testing with the TMD and DPOAE in the lying, sitting, standing, and head-down tilt (10 degrees) position. In addition, testing will be performed during sleep, when normal fluctuations of ICP occur.

Diagnostic decisions will be based on the standard invasive ICP monitoring only, and not based on the noninvasive ICP monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of suspected symptomatic hydrocephalus or idiopathic intracranial hypertension (pseudotumor cerebri)
* ICP monitoring via 25-ga needle in an existing shunt reservoir or ICP monitoring via spinal catheter has been recommended on the basis of standard clinical criteria
* Capable of providing valid signed informed consent
* Normal middle-ear function as determined by tympanometry
* DPOAE meet criteria that are required for the research
* Acoustic stapedial reflex meets criteria that are required for the research
* Subject is willing and able to return for the study

Exclusion Criteria:

* Subject is pregnant
* Subject lacks decision-making capacity
* Subject is unwilling or unable to return for the study
* Prior middle-ear disease or surgery, with the exception of tympanostomy tubes that have been removed and are healed
* Participating in the study would significantly delay or interfere with the subject's healthcare
* Subject has excess ear wax that cannot be removed safely and could potentially be pushed onto the ear drum by the insertion of the ear plugs needed for the testing
* The TMD or DPOAE do not respond to a change in posture from lying flat to standing up, which means that the anatomic connection between the inner ear and the CSF is absent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Noninvasive ICP | Day 1 (Concurrent with invasive ICP monitoring)
  Bland-Altman analysis: the difference between the noninvasive ICP and the invasive ICP is plotted against the mean of both the noninvasive and invasive ICP at each ICP level

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Williams, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States